CLINICAL TRIAL: NCT04137094
Title: Development and Pilot Testing of a Persuasive Health Communication Intervention for Emergency Department Patients Who Decline Rapid HIV/ HCV Screening
Brief Title: Development and Pilot Testing of a PHCI for Emergency Department Patients Who Decline Rapid HIV/ HCV Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1301303
Record Dates: First submitted 2019-10-16; First posted 2019-10-23 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2020-11

CONDITIONS: Hiv; Hepatitis C
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Hepatitis C

STUDY DESIGN:
Intervention Model Description: Adult ED patients who decline rapid HIV/HCV screening will be randomly assigned to the ED medical staff arm or the HIV/HCV counselor arm. Within each arm, participants further will be randomly assigned to receive the persuasive health communication intervention or watch the CDC HIV/HCV testing brochures-based video.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PHCI with HIV/HCV counselor (Experimental): A persuasive health communication intervention will be performed by a community HIV/HCV test counselor
  Interventions: Behavioral: Persuasive Health Communication Intervention
- PHCI with ED Medical Staff (Experimental): A persuasive health communication intervention will be performed by ED medical staff
  Interventions: Behavioral: Persuasive Health Communication Intervention

INTERVENTIONS:
Behavioral: Persuasive Health Communication Intervention — A persuasive health communication intervention will be performed

SUMMARY:
The Centers for Disease Control and Prevention (CDC) recommends that emergency departments (EDs) and other health care facilities conduct HIV and HCV screening to identify and link to care those with undiagnosed infections. Screening for both infections in EDs is preferable due to: the shared overlap of some risk behaviors for HIV and HCV acquisition (e.g., drug use) the relatively high co-occurrence of these infections in some populations the more complex medical needs and worse sequelae for those co-infected, and efficiency. Although some EDs have experimented with dual HIV and HCV screening, best practices on how to conduct screening so as to maximize patient screening uptake have yet to be identified.

In this pilot RCT, the investigators will examine the efficacy of the persuasive health communication intervention in convincing adult ED patients who decline rapid HIV/HCV screening to be tested for these infections. Adult ED patients who decline rapid HIV/HCV screening will be randomly assigned to the ED medical staff arm or the HIV/HCV counselor arm. Within each arm, participants further will be randomly assigned to receive the persuasive health communication intervention or to watch a CDC HIV/HCV testing brochures-based video. Following the intervention or control condition, all participants will be offered rapid HIV/HCV testing again.

DETAILED DESCRIPTION:
The investigators will conduct this R34 project at the Rhode Island Hospital ED, the primary site for many of the research team's previous HIV (Human Immunodeficiency Virus) and HCV (Hepatitis C Virus) testing studies. Dr. Beaudoin (PI) is an attending physician at the Rhode Island Hospital ED. Our multi-disciplinary team consists of researchers with extensive experience in HIV and HCV testing research, intervention development and testing, and qualitative, quantitative and cost-effectiveness research.

First, the investigators will examine our primary objective in this R34 pilot RCT( Randomized Controlled Trial) of comparing the persuasive health communication intervention to the video. Second, the investigators can compare WITHIN study arms (HIV/HCV counselor arm, ED medical staff arm) and ACROSS these study arms uptake of HIV/HCV testing among participants. Second, the design permits the investigators to obtain initial efficacy data of the persuasive health communication intervention when used by HIV/HCV counselors vs. ED medical staff (ACROSS study arms), as well as compared to the video (WITHIN study arms). Third, the design replicates our subsequent R01 RCT when the investigators compare HIV/HCV screening uptake when conducted solely by HIV/HCV counselors vs. ED medical staff.

ELIGIBILITY:
Inclusion Criteria:

* 18-64 years old
* English or Spanish speaking

Exclusion Criteria:

* HIV positive; HCV positive In an HIV vaccine trial
* On HIV pre-exposure prophylaxis medication
* In an HIV or HCV testing study
* Tested for HIV AND HCV within the past year (per EMR(Electronic Medical Record) review and patient report)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
HIV/HCV testing uptake | 10 minutes
  HIV/HCV testing will be remeasured via questionnaire following the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No